CLINICAL TRIAL: NCT02600949
Title: Pilot Study of the Feasibility and Safety of a Personalized Peptide Vaccine in Patients With Advanced Pancreatic Ductal Adenocarcinoma or Colorectal Adenocarcinoma
Brief Title: Personalized Peptide Vaccine in Treating Patients With Advanced Pancreatic Cancer or Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1029; NCI-2016-00015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-1029 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IV Pancreatic Cancer AJCC v6 and v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Imiquimod; pembrolizumab; sotigalimab; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (personalized vaccine, imiquimod) (Experimental): Patients receive personalized synthetic tumor-associated peptide vaccine therapy SC on day 1 of weeks 0, 1, 3, 4, 6, 12, and 24. Beginning 15 minutes after each vaccine is administered, patients then receive imiquimod cream topically in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI scans at baseline and at weeks 0 and 6, then every 3 months, and at week 39.
  Interventions: Drug: Imiquimod; Biological: Synthetic Tumor-Associated Peptide Vaccine Therapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Cohort B (personalized vaccine, imiquimod, pembrolizumab) (Experimental): Patients receive personalized synthetic tumor-associated peptide vaccine therapy SC on day 1 of weeks 0, 1, 3, 4, 6, 12, and 24. Beginning 15 minutes after each vaccine is administered, patients receive imiquimod cream topically. Patients also receive pembrolizumab IV over 30 minutes every 3 weeks until week 24 in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI scans at baseline and at weeks 0 and 6, then every 3 months, and at week 39.
  Interventions: Drug: Imiquimod; Biological: Pembrolizumab; Biological: Synthetic Tumor-Associated Peptide Vaccine Therapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Cohort C and D (vaccine, imiquimod, pembrolizumab, APX005M) (Experimental): Patients receive personalized synthetic tumor-associated peptide vaccine therapy SC on day 1 of weeks 0, 1, 3, 4, 6, 9, 12, 15, 18, 21, and 24. Beginning 15 minutes after each vaccine is administered, patients receive imiquimod cream topically. Patients also receive pembrolizumab IV over 30 minutes every 3 weeks until week 24 in the absence of disease progression or unacceptable toxicity. Beginning about 1 hour after each vaccine, patients also receive sotigalimab IV over 60 minutes on day 1 of weeks 0, 1, 3, 4, 6, 12, and 24 in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI scans at baseline and weeks 6,12, and 24, then every 3 months, and at week 39.
  Interventions: Drug: Imiquimod; Biological: Pembrolizumab; Biological: Sotigalimab; Biological: Synthetic Tumor-Associated Peptide Vaccine Therapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Imiquimod — Applied topically
  Other Names: Aldara; R 837; S 26308; Zyclara
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Cohort B (personalized vaccine, imiquimod, pembrolizumab); Cohort C and D (vaccine, imiquimod, pembrolizumab, APX005M)
Biological: Sotigalimab — Given IV
  Other Names: APX 005; APX 005M; APX-005M; APX005M; CD40 Agonistic Monoclonal Antibody APX005M; EPI-0050
  Arms: Cohort C and D (vaccine, imiquimod, pembrolizumab, APX005M)
Biological: Synthetic Tumor-Associated Peptide Vaccine Therapy — Given SC
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; CT
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MR; MRI Scan; Nuclear Magnetic Resonance Imaging; NMR; NMRI; NMR Imaging

SUMMARY:
This phase I trial studies the side effects and best way to give personalized peptide vaccine in patients with pancreatic or colorectal cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Personalized peptide vaccine is a vaccine developed from patient's own tumor cells and blood in order to use as a biological therapy. Biological therapies, such as personalized peptide vaccine may attack tumor cells and stop them from growing or kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate that developing a custom vaccine for metastatic pancreatic ductal adenocarcinoma (PDA) and colorectal cancer (CRC) patients is feasible. (cohorts A and B)

II. Show that a custom peptide-based vaccine in combination with imiquiomod, pembrolizumab, and/or sotigalimab (APX005M) is safe. (cohorts A and B and C and D)

SECONDARY OBJECTIVES:

I. Determine the clinical benefit of the peptide vaccine alone or combined with pembrolizumab or pembrolizumab and APX005M. (cohorts A and B and C and D)

II. Demonstrate the antigenicity of each vaccine. (cohorts A and B and C and D)

III. The change in neoantigen-specific T cell responses at 12 weeks after initiation of personalized peptide vaccination. (cohorts C and D)

IV. Relapse-free survival and circulating tumor deoxyribonucleic acid (ctDNA) clearance rate. (cohorts C and D)

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT A: Patients receive personalized synthetic tumor-associated peptide vaccine therapy subcutaneously (SC) on day 1 of weeks 0, 1, 3, 4, 6, 12, and 24. Beginning 15 minutes after each vaccine is administered, patients then receive imiquimod cream topically in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) scans at baseline and at weeks 0 and 6, then every 3 months, and at week 39.

COHORT B: Patients receive personalized synthetic tumor-associated peptide vaccine therapy SC on day 1 of weeks 0, 1, 3, 4, 6, 12, and 24. Beginning 15 minutes after each vaccine is administered, patients receive imiquimod cream topically. Patients also receive pembrolizumab intravenously (IV) over 30 minutes every 3 weeks until week 24 in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI scans at baseline and at weeks 0 and 6, then every 3 months, and at week 39.

COHORTS C AND D: Patients receive personalized synthetic tumor-associated peptide vaccine therapy SC on day 1 of weeks 0, 1, 3, 4, 6, 9, 12, 15, 18, 21, and 24. Beginning 15 minutes after each vaccine is administered, patients receive imiquimod cream topically. Patients also receive pembrolizumab IV over 30 minutes every 3 weeks until week 24 in the absence of disease progression or unacceptable toxicity. Beginning about 1 hour after each vaccine, patients also receive sotigalimab IV over 60 minutes on day 1 of weeks 0, 1, 3, 4, 6, 9, 12, 15, 18, 21, and 24 in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI scans at baseline and weeks 6,12, and 24, then every 3 months, and at week 39.

After completion of study treatment, patients are followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic CRC or PDA planned to or have undergone complete surgical resection (metastatectomy) and also for PDA participants with localized disease planned for primary tumor resection.
* Any lines (including zero) of therapy prior to tissue harvest.
* Adequate tumor tissue availability
* Adults (age ≥ 18)
* ECOG PS 0-1
* Life expectancy >12 months for Cohort C and >9 months for Cohort D
* Adequate organ and marrow function
* Ability to understand and the willingness to sign a written informed consent document.
* As the effects of a peptide based vaccine, pembrolizumab or APX005M on the developing human fetus are unknown, women of child-bearing potential and men must agree to use adequate contraception at study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant, she should inform her treating physician immediately. Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), sexually active participants must use birth control during and for >120 days after the study. Abstinence is also an acceptable form of birth control.
* For Cohort C only: participants must have metastatic CRC and are planned to or have undergone complete metastecomy/ies and agree to have post-operative blood draw for ctDNA testing within 6 weeks following surgical resection.

Exclusion Criteria:

* History of HIV or AIDS
* Patients with brain metastasis
* Serious autoimmune conditions
* Use of chronic immune suppressive medications.
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women of child bearing potential who are pregnant or breastfeeding. Women with a positive pregnancy test at enrollment or prior to administration of vaccine. .
* Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to therapy drugs or their components.
* Has a known additional malignancy that is progressing or requires active treatment.
* Active coagulopathy.
* History of arterial thrombosis within 3 months prior to starting study treatment.
* History of New York Heart Association Class 3-4 heart failure or myocardial infarction within 6 months prior to starting therapy.
* Known history of Hepatitis B or known active Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of enrolled patients for whom a personalized vaccine is developed and ready to administer (cohorts A and B) | Up to 12 weeks post-enrollment
Proportion of enrolled patients who receive at least 1 dose of vaccine at any time post-enrollment (cohorts A and B) | Up to 44 weeks
Incidence of adverse events (AEs) | Up to 24 weeks
  Defined as the proportion of subjects who experience at least one toxicity event per National Cancer Institute Common Toxicity Criteria for Adverse Events version 4.0. A toxicity event is defined as at least one grade 3 or 4 non-hematologic or grade 4 hematologic toxicity. Proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval.

SECONDARY OUTCOMES:
Proportion of patients who have received at least one dose of vaccine that is alive and progression free defined based on response criteria according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | At 12 weeks post-vaccination (second re-staging scan)
  Progression free includes complete response (CR), partial response (PR), and stable disease (SD). The target proportion is 45%, and a proportion of 20% or lower will be considered as not having the desired efficacy.
Progression-free survival (cohorts A and B and C) | The time between the date of first vaccination and evidence of progression on computed tomography scan or the date of death due to any cause, assessed up to 6 months after the last dose of vaccine
  Estimated by the Kaplan-Meier method, along with the 95% confidence intervals, and log-rank test will be used to assess the time to event variable differences under different patient subgroups.
Response rate (cohort A and B) | Up to 12 weeks
  Response rate includes both CR and PR and will be evaluated using a Simon optimal two-stage design.
Change in tumor biomarker (CA19-9, carcinoembryonic antigen [CEA] or circulating free deoxyribonucleic acid [cfDNA] mutation) | Up to 6 months
Overall survival | The time from first vaccination to death, assessed up to 6 months after the last dose of vaccine
  Estimated by the Kaplan-Meier method, along with the 95% confidence intervals, and log-rank test will be used to assess the time to event variable differences under different patient subgroups.
Recurrence-free survival (cohort C and D) | Up to 6 months
  Estimated by the Kaplan-Meier method.
Rate of circulating deoxyribonucleic acid (ctDNA) clearance (cohort C and D) | Up to 6 months
  A linear mixed model will also be fitted to correlate ctDNA clearance and neoantigen-specific CD8+ T cell over time.
Change in neoantigen-specific T cell response (cohort C and D) | Baseline to 12 weeks after initiation of personalized peptide vaccination
  The difference in log2 transformed T cell response from baseline to 12 weeks will be calculated for each peptide and patient. This endpoint will focus upon the log2-fold change at 12 weeks for the max peptide (i.e., the peptide with the greatest change). Descriptive statistics, including mean, standard deviation, median and range, will be used to summarize the changes. A paired t-test will be used to evaluate the changes from baseline to 12 weeks post initiation of vaccination.
Correlation of T-cell activation against vaccinated peptides and ctDNA dynamics (cohort C and D) | Up to 6 months
Tumor microenvironment immune infiltration and progression biopsies (cohort C and D) | Baseline, up to 6 months
T cell IFN-gamma release in response to selected personalized peptide antigens | Up to 6 months
Levels of intracellular cytokine staining of T cells | Up to 6 months
  Assessed by flow cytometry in response to stimulation with personalized peptide antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Overman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org